CLINICAL TRIAL: NCT01876979
Title: Erich Arch Bars vs. IMF Screws for Placement of Maxillomandibular Fixation: Which is More Time Effective in the Operating Room Setting?
Brief Title: Arch Bars vs. IMF (Intermaxillary Fixation) Screws: Cost Effectiveness Based on Time Duration of Device Placement.
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Extended study duration
Sponsor: Christiana Care Health Services (Other)
Responsible Party: Principal Investigator, Daniel Meara, Oral and Maxillofacial Surgery Resident, Christiana Care Health Services
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CCC# 33082; DDD# 602252 (Other: ChristianaCHS)
Record Dates: First submitted 2013-06-11; First posted 2013-06-13 (Estimated); Results first posted 2017-06-28 (Actual); Last update posted 2017-06-28 (Actual); Status verified 2017-05

CONDITIONS: Mandible Fracture
MeSH Terms: conditions — Mandibular Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- IMF Screws (Active Comparator): Use of IMF screws as a means to wire the jaws.
  Interventions: Device: IMF Screws
- Erich Arch Bars (Active Comparator): Use of Erich Arch bars in the wiring of the jaws.
  Interventions: Device: Erich Arch Bars

INTERVENTIONS:
Device: IMF Screws — stainless steel screws placed in bone
  Other Names: Synthes IMF screws
  Arms: IMF Screws
Device: Erich Arch Bars — Surgical braces wired around teeth
  Arms: Erich Arch Bars

SUMMARY:
Determining the cost effectiveness, based on the time duration of application, of two methods of wiring the jaws together during surgery to repair mandible fractures. One technique is more expensive but faster in application, while the other is less expensive and takes more time to apply.

DETAILED DESCRIPTION:
Purpose:

To identify which option of wiring the jaws together during treatment of mandible fractures is more cost effective to the patient, Erich arch bars or IMF (Intermaxillary Fixation) screws. Patients who sustain mandible fractures that meet the inclusion criteria will be randomized to one of the two treatment types listed above. The overall treatment in both categories is consistent with the standard of care, the only difference being the method utilized to achieve intermaxillary fixation during the course of the surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-70
* Patients with no greater than one (1) open fracture of the tooth-bearing mandible
* Mandibular angle fractures ± Ramus or subcondylar fracture
* Body/symphysis ± subcondylar
* Isolated angle fracture
* Isolate subcondylar fractures
* Bilateral subcondylar fractures
* Any condylar head/neck fracture requiring treatment
* Patients who are candidates for treatment of their fractures in the operating room setting

Exclusion Criteria:

* Patients younger than 18 or older than 70
* Patients with developing tooth buds anterior to the second molars
* Patients with inadequate stability of occlusion
* Edentulism
* Unstable vertical and horizontal stops to the occlusion
* Patients with disorders affecting bone healing, metabolism and turnover
* Those patients on bisphosphonates, oral or IV
* Patients with evidence of intrabony pathology of the mandible or maxilla
* The presence of any of the following:
* Greater than one (1) open fracture of the tooth-bearing mandible
* Bilateral angle fractures are exempt from this
* Comminuted fractures of the mandible
* Concomitant infection, or osteomyelitis of the mandible
* Mechanism of injury
* Pathologic fracture
* Gun-shot wounds

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2013-07; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Meara, MD, Principal Investigator — Christiana Care Health Services; Daniel J Meara, MS, MD, DMD, Study Chair — Christiana Care Health Services
Locations (2):
- United States (2):
  - Christiana Care Hospital, Newark, Delaware
  - Wilmington Hospital, Wilmington, Delaware

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | IMF Screws | Erich Arch Bars
Started | 2 | 3
Completed | 0 | 0
Not Completed | 2 | 3
Not completed — Physician Decision | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Intermaxillary Fixation Screws: Use of Intermaxillary Fixation screws as a means to wire the jaws.
  IMF Screws: stainless steel screws placed in bone
- Total: Total of all reporting groups
Arm/Group | Intermaxillary Fixation Screws | Erich Arch Bars | Total
Number analyzed (Participants) | 2 | 3 | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 3 | 5
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 2 | 3 | 5
Duration to Maxillomandibular Fixation (minutes) [Mean (Full Range); unit: minutes] | 17 [11 to 23] | 40.3 [35 to 50] | 28.7 [11 to 50]

OUTCOME MEASURES:

1. Primary Outcome: Time
Description: Time duration for the application of device, in minutes.
Time Frame: Time duration of placement of device in operating room
Measure: Mean (Full Range); unit: minutes
Arm/Group | IMF Screws | Erich Arch Bars
Number analyzed (Participants) | 2 | 3
minutes | 17 [11 to 23] | 40.3 [35 to 50]

ADVERSE EVENTS:
Arm/Group | IMF Screws | Erich Arch Bars
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/3
Other Adverse Events (participants affected / at risk) | 0/2 | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes